CLINICAL TRIAL: NCT03402087
Title: An Open-Label, Single-Sequence Study to Investigate the Effects of BMS-986165 on the Single-Dose Pharmacokinetics of Methotrexate in Healthy Male Subjects
Brief Title: A Study to Investigate BMS-986165 and Methotrexate in Healthy Male Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-025; 2017-004177-13 (EudraCT Number)
Record Dates: First submitted 2018-01-05; First posted 2018-01-18 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Lupus; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate; Leucovorin; deucravacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BMS-986165+Methotrexate+Leucovorin (Experimental): Three treatments administered
  Interventions: Drug: Methotrexate; Drug: Leucovorin; Drug: BMS-986165

INTERVENTIONS:
Drug: Methotrexate — Specified dose on specified days
  Other Names: MTX
Drug: Leucovorin — Specified dose on specified days
  Other Names: LEU
Drug: BMS-986165 — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate effects of BMS-986165 on blood levels of methotrexate given as a single dose in healthy male patients.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body Mass Index (BMI): 18.0 - 32.0 kg/m2
* Normal renal function at screening

Exclusion Criteria:

* Any medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, liver disease
* Any contraindication indicated in the MTX package insert
* History or presence of chronic bacterial or viral infection
* History or presence of an autoimmune disorder
* Any significant acute or chronic medical illness
* Active TB requiring treatment or documented latent TB within the previous 3 years
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect absorption

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Approximately 14 days
Time to attain maximum observed plasma concentration (Tmax) | Approximately 14 days
Area under the plasma concentration-time curve up to time T, where T is the last point with concentrations above the lower limit of quantitation [AUC(0-T)] | Approximately 14 days
Area under the plasma concentration-time curve from time 0 to infinity [AUC(INF)] | Approximately 14 days
Terminal elimination rate constant (kel) | Approximately 14 days
Terminal elimination half life, calculated as 0.693/kel (T-HALF) | Approximately 14 days
Apparent oral clearance (CL/F) | Approximately 14 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Approximately 19 days
Incidence of serious adverse events (SAEs) | Approximately 19 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx